CLINICAL TRIAL: NCT02564263
Title: A Phase III Randomized Open-Label Study of Single Agent Pembrolizumab vs Physicians' Choice of Single Agent Docetaxel, Paclitaxel, or Irinotecan in Subjects With Advanced/Metastatic Adenocarcinoma and Squamous Cell Carcinoma of the Esophagus That Have Progressed After First-Line Standard Therapy (KEYNOTE-181)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Investigator's Choice Standard Therapy for Participants With Advanced Esophageal/ Esophagogastric Junction Carcinoma That Progressed After First-Line Therapy (MK-3475-181/KEYNOTE-181)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-181; 163145 (Registry Identifier: JAPAN-CTI); MK-3475-181 (Other: Merck); KEYNOTE-181 (Other: Merck); 2015-002782-32 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Carcinoma; Esophagogastric Junction Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Death-Ligand 2 (PDL2, PD-L2); Gene expression profiling (GEP)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants received pembrolizumab 200 mg, intravenously (IV) on Day 1 of every 21-day (3-week) cycle for up to 35 administrations (up to approximately 25 months).
  Interventions: Biological: pembrolizumab
- Chemotherapy (Active Comparator): Participants received Investigator's choice of paclitaxel 80-100 mg/m^2 IV on Days 1, 8, and 15 of every 28-day (4-week) cycle, OR docetaxel 75 mg/m^2 IV on Day 1 of every 21-day (3-week) cycle, OR irinotecan 180 mg/m^2 IV on Day 1 of every 14-day (2-week) cycle (up to approximately 19 months).
  Interventions: Drug: paclitaxel; Drug: docetaxel; Drug: irinotecan

INTERVENTIONS:
Biological: pembrolizumab — 200 mg administered as IV infusion on Day 1 of every 21-day cycle
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: paclitaxel — 80-100 mg/m^2 administered as IV infusion on Days 1, 8, and 15 of each 28-day cycle
  Other Names: TAXOL®
  Arms: Chemotherapy
Drug: docetaxel — 75 mg/m^2 administered as IV infusion on Day 1 of every 21-day cycle
  Other Names: TAXOTERE®
  Arms: Chemotherapy
Drug: irinotecan — 180 mg/m^2 administered as IV infusion on Day 1 of every 14-day cycle
  Other Names: CAMPTOSAR®
  Arms: Chemotherapy

SUMMARY:
In this study, participants with advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or Siewert type I adenocarcinoma of the esophagogastric junction (EGJ) that had progressed after first-line standard therapy were randomized to receive either pembrolizumab (MK-3475) OR the Investigator's choice of standard chemotherapy with paclitaxel, docetaxel, or irinotecan.

The primary study hypothesis was that treatment with pembrolizumab would prolong overall survival (OS) as compared to treatment with standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of adenocarcinoma or squamous cell carcinoma of the esophagus or Siewert type I adenocarcinoma of the EGJ
* Metastatic disease or locally advanced, unresectable disease
* Life expectancy of greater than 3 months
* Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Documented radiographic or clinical disease progression on no more or less than one previous line of standard therapy
* Can provide either a newly obtained or archival tumor tissue sample for intra-tumoral immune-related testing and for anti-programmed cell death (PD)-1
* Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel, docetaxel or irinotecan
* Adequate organ function

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment
* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis (includes past history or current metastasis)
* Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent
* Has had a severe hypersensitivity reaction to treatment with another mAb
* Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1), or anti-PD-L2 agent, or previously participated in Merck pembrolizumab (MK-3475) study
* Has a known additional malignancy that has progressed or required active treatment within the last 5 years with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers, and in-situ or intra-mucosal pharyngeal cancer
* Received a live vaccine within 30 days of the first dose of study treatment
* Known history of human immunodeficiency virus (HIV) infection
* Known history of or is positive for hepatitis B or known active hepatitis C
* History of non-infectious pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study starting with the screening visit through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel, docetaxel or irinotecan
* Known allergy, hypersensitivity, or contraindication to paclitaxel, docetaxel, or irinotecan or any components used in their preparation
* Experienced weight loss >10% over approximately 2 months prior to first dose of study treatment
* Has ascites or pleural effusion by physical exam
* Has experienced documented objective radiographic or clinical disease progression during or after receiving >1 line of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Derived] Adenis A, Kulkarni AS, Girotto GC, de la Fouchardiere C, Senellart H, van Laarhoven HWM, Mansoor W, Al-Rajabi R, Norquist J, Amonkar M, Suryawanshi S, Bhagia P, Metges JP. Impact of Pembrolizumab Versus Chemotherapy as Second-Line Therapy for Advanced Esophageal Cancer on Health-Related Quality of Life in KEYNOTE-181. J Clin Oncol. 2022 Feb 1;40(4):382-391. doi: 10.1200/JCO.21.00601. Epub 2021 Nov 3. PMID 34730989
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the time of the primary analysis data cut-off of 15-Oct-2018, 67 participants were ongoing in the study.
Period: Overall Study
Arm/Group | Pembrolizumab | Chemotherapy
Started | 314 | 314
Treated | 314 | 296
Received Second Course of Pembrolizumab | 5 | 0
Completed | 0 | 0
Not Completed | 314 | 314
Not completed — Adverse Event | 31 | 29
Not completed — Death | 270 | 262
Not completed — Withdrawal by Subject | 4 | 19
Not completed — Sponsor's decision | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg IV on Day 1 of every 21-day (3-week) cycle for up to 35 administrations (up to approximately 25 months).
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Chemotherapy | Total
Number analyzed (Participants) | 314 | 314 | 628
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (9.4) | 62.0 (9.6) | 62.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 273 | 271 | 544
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 25 | 44
  Not Hispanic or Latino | 288 | 273 | 561
  Unknown or Not Reported | 7 | 16 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 126 | 122 | 248
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 179 | 172 | 351
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 4 | 11 | 15
Programmed Death-Ligand 1 (PD-L1) Status: Combined Positive Score (CPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression levels by immunohistochemistry assay on tumor tissue from a newly obtained biopsy. PD-L1 CPS was calculated as the number of PD-L1 positive cells (tumor cells, macrophages, lymphocytes) divided by the total tumor cells and is expressed as a percentage. Participants were classified based on their PD-L1 tumor status as being either PD-L1 CPS ≥10 or PD-L1 CPS <10.
  Participants
    PD-L1 CPS ≥10 | 109 | 117 | 226
    PD-L1 CPS <10 | 199 | 194 | 393
    Not Evaluable | 6 | 3 | 9
Geographic Region [Count of Participants; unit: Participants] — Participants were classified based on their geographic region of enrollment as either being from Asia or from outside of Asia (Rest of World [RoW]).
  Participants
    Asia | 121 | 122 | 243
    RoW | 193 | 192 | 385
Tumor Histology [Count of Participants; unit: Participants] — Participants were classified based on their tumor histology (cell type) as either having squamous cell carcinoma or having adenocarcinoma of esophagus and esophagogastric junction (EGJ) Siewert type I.
  Participants
    Squamous cell carcinoma | 199 | 204 | 403
    Adenocarcinoma of esophagus & EGJ Siewert type I | 115 | 110 | 225

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: OS was defined as the time from randomization to death due to any cause. Median OS in participants with SCC of the esophagus is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: The efficacy analysis population consisted of all randomized participants with SCC of the esophagus. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 198 | 203
Months | 8.2 [6.7 to 10.3] | 7.1 [6.1 to 8.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.00894, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.63 to 0.96] — Cox regression model with treatment as a covariate stratified by geographic region (Asia vs RoW)

2. Primary Outcome: Overall Survival (OS) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: OS was defined as the time from randomization to death due to any cause. Median OS in participants with a PD-L1 CPS ≥10 is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: The efficacy analysis population consisted of all randomized participants with a PD-L1 CPS ≥10. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 107 | 115
Months | 9.3 [6.6 to 12.5] | 6.7 [5.1 to 8.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.00855, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.52 to 0.94] — Cox regression model with treatment as a covariate stratified by geographic region (Asia vs RoW) & tumor histology (SCC vs adenocarcinoma/Siewert type 1 adenocarcinoma of the esophagogastric junction [EGJ])

3. Primary Outcome: Overall Survival (OS) in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Median OS in all participants is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: The efficacy analysis population consisted of all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 314 | 314
Months | 7.1 [6.2 to 8.1] | 7.1 [6.3 to 8.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0531, Log Rank — One-sided p-value based on stratified maximum weighted log rank test: the maximum of the log-rank test statistic & a weighted log-rank Fleming-Harrington (0,1) test statistic; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.75 to 1.05] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS as assessed by blinded independent central review per RECIST 1.1 in all participants is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 314 | 314
Months | 2.1 [2.1 to 2.2] | 3.4 [2.8 to 3.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.287, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.94 to 1.31] — Cox regression model with treatment as a covariate stratified by geographic region (Asia vs RoW) & tumor histology (SCC vs adenocarcinoma/Siewert type 1 adenocarcinoma of the EGJ)

5. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of all participants who experienced a CR or PR is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 314 | 314
Percentage of Participants | 13.1 [9.5 to 17.3] | 6.7 [4.2 to 10.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0037, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0 versus; H1: difference in %>0; Difference in Percentages = 6.4, 95% CI 2-sided [1.7 to 11.2] — Miettinen & Nurminen method stratified by geographic region (Asia vs RoW) & tumor histology (SCC vs adenocarcinoma/Siewert type I adenocarcinoma of the EGJ)

6. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS as assessed by blinded independent central review per RECIST 1.1 is presented for participants with SCC of the esophagus.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 198 | 203
Months | 2.2 [2.1 to 3.2] | 3.1 [2.2 to 3.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.216, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.13] — Cox regression model with treatment as a covariate stratified by geographic region (Asia vs RoW)

7. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS as assessed by blinded independent central review per RECIST 1.1 is presented for participants with a PD-L1 CPS ≥10.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 107 | 115
Months | 2.6 [2.1 to 4.1] | 3.0 [2.1 to 3.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.015, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.54 to 0.97] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants with SCC of the esophagus who experienced a CR or PR is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 198 | 203
Percentage of Participants | 16.7 [11.8 to 22.6] | 7.4 [4.2 to 11.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0022, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0; H1: difference in %>0; Difference in Percentages = 9.2, 95% CI 2-sided [3.0 to 15.8] — Miettinen & Nurminen method stratified by geographic region (Asia vs RoW)

9. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants with a PD-L1 CPS ≥10 who experienced a CR or PR is presented.
Time Frame: Through Final Analysis data cutoff date of 15-Oct-2018 (up to approximately 34 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 107 | 115
Percentage of Participants | 21.5 [14.1 to 30.5] | 6.1 [2.5 to 12.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0006, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0; H1: difference in %>0; Difference in Percentages = 15.1, 95% CI 2-sided [6.2 to 24.7] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who experienced ≥1 AE is presented.
Time Frame: Through End-of-Trial Analysis data cutoff date of 14-Mar-2022 (up to approximately 6 years)
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 314 | 296
Participants | 301 | 288

11. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Through End-of-Trial Analysis data cutoff date of 14-Mar-2022 (up to approximately 6 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 314 | 296
Participants | 40 | 42

ADVERSE EVENTS:
Time Frame: Through End-of-Trial Analysis data cutoff date of 14-Mar-2022 (up to approximately 6 years)
Description: All-Cause Mortality (ACM) was reported for all randomized participants. Five participants got a second course of pembrolizumab and were monitored for AEs and ACM. Safety was analyzed in participants who got ≥1 dose of study drug. Per protocol, disease progression of cancer was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to study drug are excluded as AEs.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg, intravenously (IV) on Day 1 of every 21-day (3-week) cycle for up to 35 administrations (up to approximately 25 months).
- Pembrolizumab Second Course: Qualified participants who received pembrolizumab as a first course and stopped the first course of pembrolizumab due to complete response (CR) or completed the first course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
Arm/Group | Pembrolizumab First Course | Chemotherapy | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 305/314 | 305/314 | 3/5
Serious Adverse Events (participants affected / at risk) | 127/314 | 121/296 | 1/5
Other Adverse Events (participants affected / at risk) | 285/314 | 281/296 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=314) | Chemotherapy (N=296) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 22 (24) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 11 (12) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 10 (10) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 4 (4) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (15) | 22 (26) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 12 (13) | 5 (5) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (4) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=314) | Chemotherapy (N=296) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 52 (60) | 83 (110) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 36 (65) | 0 (0)
Hypothyroidism (Endocrine disorders) | 37 (40) | 7 (7) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 34 (36) | 27 (32) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16) | 17 (19) | 0 (0)
Constipation (Gastrointestinal disorders) | 56 (63) | 56 (63) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 38 (65) | 79 (120) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 11 (13) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 40 (44) | 26 (27) | 1 (1)
Nausea (Gastrointestinal disorders) | 59 (66) | 83 (110) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 28 (30) | 0 (0)
Vomiting (Gastrointestinal disorders) | 37 (45) | 53 (74) | 0 (0)
Asthenia (General disorders) | 45 (48) | 43 (58) | 0 (0)
Fatigue (General disorders) | 67 (70) | 87 (121) | 0 (0)
Malaise (General disorders) | 15 (18) | 19 (26) | 0 (0)
Oedema peripheral (General disorders) | 19 (20) | 19 (19) | 0 (0)
Pyrexia (General disorders) | 31 (41) | 45 (58) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (17) | 13 (15) | 1 (2)
Alanine aminotransferase increased (Investigations) | 22 (26) | 10 (16) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 26 (33) | 14 (16) | 1 (1)
Blood creatinine increased (Investigations) | 8 (11) | 3 (4) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 3 (4) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (10) | 9 (15) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 50 (113) | 0 (0)
Weight decreased (Investigations) | 39 (39) | 34 (43) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 52 (114) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 76 (82) | 76 (97) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (21) | 14 (14) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (13) | 6 (7) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (23) | 15 (16) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (15) | 29 (40) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (27) | 17 (24) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (26) | 19 (22) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 38 (40) | 24 (27) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 25 (31) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (9) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 6 (7) | 25 (28) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 52 (53) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (25) | 16 (42) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (46) | 30 (33) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 17 (21) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 88 (88) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (27) | 8 (8) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 20 (24) | 25 (27) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02564263/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02564263/SAP_002.pdf